CLINICAL TRIAL: NCT07261878
Title: Injectable Platelet Rich Fibrin (I-PRF) With Xenograft in Intrabony Defects of Periodontitis Patient Stage III Versus Xenograft Alone
Brief Title: Treatment of Intrabony Defect in Patient With Periodontitis Stage III by Using I-PRF and Xenograft
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ola Alsareh, Oral Medicine, Periodontology, Oral Diagnosis and Radiology Department Faculty of Dental Medicine for Girls Al-Azhar University, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-ME-24-05
Record Dates: First submitted 2025-08-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Intrabony Defect; Intrabony Defects in Chronic Periodontitis
Keywords: I-PRF with xenograft
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- injectable platelet rich fibrin and xenograft (Other): Intrasulcular incisions will be performed buccally and lingually/palatally on the affected tooth and extended one adjacent tooth mesially and distally, using 15c blades. Following mucoperiosteal flap elevation, thorough debridement will be performed using ultrasonic scalers and curettes until defects are clear from any granulation tissue, and the defect morphology will be visually explored and recorded .In the group 2: xenograft (Bovin xenograft) with injectable platelet Rich fibrin (I- PRF) will be applied to the intrabony defect area.
  Interventions: Procedure: injectable platelet rich fibrin and xenograft; Procedure: Xenograft alone
- xenograft alone (Active Comparator): Intrasulcular incisions will be performed buccally and lingually/palatally on the affected tooth and extended one adjacent tooth mesially and distally, using 15c blades. Following mucoperiosteal flap elevation, thorough debridement will be performed using ultrasonic scalers and curettes until defects are clear from any granulation tissue, and the defect morphology will be visually explored and recorded, inserting the xenograft to the defect
  Interventions: Procedure: injectable platelet rich fibrin and xenograft; Procedure: Xenograft alone

INTERVENTIONS:
Procedure: injectable platelet rich fibrin and xenograft — Elevation of papilla preservation flap at the site of 3mm infrabony defect ,prepearing the I-PRF which is obtained from the patients own blood , centrifuged at 700 rpm in 3 min and mixed with xenograft than placed at the defect area after removal all the granulation tissue follow up after 3 and 6 months intervals
Procedure: Xenograft alone — Elevation of papilla preservation flap at the site of 3mm infrabony defect after removal all the granulation tissue, the xenograft alone inserted to the defect, suturing and follow up after 3 and 6 months intervals

SUMMARY:
Evaluate of the injectable platelet rich fibrin (I-PRF) with xenograft in Intrabony defects of Periodontitis patient stage III versus Xenograft alone.

DETAILED DESCRIPTION:
All surgical procedures will be conducted by a single operator. Following administration of local anesthesia, intrasulcular incisions will beperformed buccally and lingually/palatally on the affected tooth and extended one adjacent tooth mesially and distally, using 15c blades. Following mucoperiosteal flap elevation, thorough debridement will be performed using ultrasonic scalers and curettes until defects are clear from any granulation tissue, and the defect morphology will be visually explored and recorded. In the group1: xenograft alone(Bovin xenograft)will be applied to the intrabony defect area. In the group 2: xenograft (Bovin xenograft) with injectable platelet Rich fibrin (I- PRF) will be applied to the intrabony defect area. Preperation of Injectable platelate Rich Fibrin (I-PRF) : will be prepared for each patient as follows: 5 ml of venous blood will be collected from the patient blood then placed in a plastic tube without any added material or coagulant and centrifuged at 700 rpm for 3 min. then mixed with Xenograft. Finally, the flap will be passively repositioned using interrupted 4-0 silk

ELIGIBILITY:
Inclusion Criteria:

1. Patient should have localized Periodontitis stage III grade B with pocket depth ≥ 6mm; indicated for periodontal surgery
2. Patient's agreement to the surgical procedure and clinical trial.
3. Age ranged between 30-55 years old.
4. Intrabony defects with depth ≥3mm.
5. Free from any systemic conditions and no previous drug affect bone metabolism

Exclusion Criteria:

1. Smoking.
2. Pregnant women.
3. Patients in variation in anatomical landmarks.
4. Patients with psychological problems.
5. Patients with abnormal habits.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
Radiographic parameters | 6 months after treatment
  • The bone fill after 6 months postoperatively using digital periapical radiography using parallel technique.

SECONDARY OUTCOMES:
Pocket depth (PD) | presurgically, 3 and 6 months interval after treatment
  will be assessed by William graduated periodontal Probe in 4 surfaces of the tooth
Plaque index (PI) | pre-surgically 3 months and 6 months respectively
  According to Silness & Loe, 4 readings will be recorded for each surface of the teeth (buccal, lingual, mesial and distal) and it is given a score from 0-3
Gingival index (GI) | pre-surgically 3 months and 6 months respectively
  presence or absence of bleeding on upon gentle probing
Clinical attachment level (CAL) | pre-surgically 3 months and 6 months respectively
  will be measured from the cement-enamel junction to the base of the pocket

CONTACTS AND LOCATIONS:
Overall Officials: Eatemad Ahmed Shoreibah A Shoreibah, Professor, Study Chair — Al-Azhar University
Locations (2):
- Egypt (2):
  - Faculty of Dental Medicine for Girls, Al- Azhar University, Cairo, Cairo Governorate
  - Ola Jamal, Cairo, Cairo Governorate

IPD SHARING:
Plan to Share IPD: Undecided